CLINICAL TRIAL: NCT06003764
Title: Efficacy of Pulsed Electromagnetic Field Therapy on Acute Radiodermatitis in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mahmoud H Mohamed, PhD, Assistant Professor of Physical Therapy, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AhramCU
Record Dates: First submitted 2023-08-12; First posted 2023-08-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dermatitis, Radiation Induced
Keywords: PEMFT, DERMATITIS, RADIOTHERAPY
MeSH Terms: conditions — Radiodermatitis; Dermatitis

STUDY DESIGN:
Intervention Model Description: randomized, single blinded controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed electromagnetic field group (Experimental): Pulsed electromagnetic
  Interventions: Other: Pulsed electromagnetic field; Other: traditional skin care
- Placebo group (Placebo Comparator): traditional skin care
  Interventions: Other: traditional skin care

INTERVENTIONS:
Other: Pulsed electromagnetic field — low-frequency PEMFT (15 Hz, 50% intensity output for 5 s/min for 20 minutes)
  Arms: Pulsed electromagnetic field group
Other: traditional skin care — traditional skin care( the patients received the institutional standard skin care, which encompassed 3×/day application of topical, hydroactive colloid gel, from the first day of RT. In case of a painful skin reaction and/or moist desquamation, a foam, absorbent, self-adhesive silicone dressing was used. Additionally, the patient was advised to follow the general skin care guidelines (e.g., no tie, no electric shaving, no aftershave, gentle washing with or without mild soap, patting dry with a soft towel instead of rubbing

SUMMARY:
This study aims to evaluate the impact of PEMF on acute radiodermatitis in breast cancer patient and post mastectomy patients.

DETAILED DESCRIPTION:
The objective is to understand the effect of PEMF on skin thickness and toxicity after radiotherapy on breast cancer.

The study included 50 adult female breast cancer undergoing whole-breast irradiation.

This is a randomized, controlled clinical trial was conducted at the outpatient clinic of the Faculty of Physical Therapy, Ahram Canadian University, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients undergoing HF-WBI post-lumpectomy with or without chemotherapy.
* Unilateral breast cancer
* Age from 35-55 years.

Exclusion Criteria:

* Patients had previous irradiation to the same breast.
* Patients had bilateral breast cancer.
* Patients had metastatic disease.
* when the use of bolus material was required to deliver RT.
* Patients had a pre-existing skin condition or open wound in the treatment area.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females with Breast cancer
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Ultrasonography skin thickness measurement. | pre treatment, every two weeks of treatment( total weeks 8 weeks) of treatment for up to 2 months total time.
  Ultrasonography was performed before radiotherapy and every two week during radiotherapy, approximately at the same time as skin toxicity assessments.
  The machine (L15-4 linear-array transducer; Supersonics Aixplorer; Supersonic Imagine; France) and settings were used for all examinations, including gain, depth and frequency. Exams are performed at room temperature of 20-25°C with the patient supine, hands raised above the head and the ultrasound scans are performed by an experienced sonographer. Standard echo gel is used as a couplant between the skin surface and the probe. To ensure good coupling of the probe/skin interface, in addition to the gel, a sound-guiding pad with a size of 130 × 120 × 10 mm was used. During all examinations, special care was taken to avoid any pressure on the skin surface, and the probe is gently applied to the surface

SECONDARY OUTCOMES:
Radiation Therapy Oncology Group (RTOG) SCALE | pre treatment, every two weeks of treatment( total weeks 8 weeks) of treatment for up to 2 months total time.
  0 No change
  1. Faint erythema or dry desquamation
  2. Moderate to brisk erythema; patchy, moist desquamation, mostly confined to skin folds and creases; moderate edema
  3. Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion
  4. Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated

CONTACTS AND LOCATIONS:
Locations (1):
- ahram canadian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed MH, Selim MN, Mohamed ME, Elmeligie MM, Kadry AM, Abdelrazik RK, Samir SM, Kamel RM, Kamal KA, Elshazly M. Efficacy of pulsed electromagnetic field therapy on acute radiodermatitis in breast cancer patients: a randomized controlled study. Support Care Cancer. 2026 Feb 5;34(3):168. doi: 10.1007/s00520-026-10322-9. PMID 41642361